CLINICAL TRIAL: NCT05373108
Title: Impact of Endothelin-1 on the Development of Cardiac Allograft Vasculopathy in Heart Transplant Recipients: Endothelin Receptor Antagonism and Vasomotor Function
Brief Title: Endothelin-1 and Cardiac Allograft Vasculopathy (CAV)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: American Heart Association (Other); Janssen, LP (Industry)
Responsible Party: Principal Investigator, Rushi V. Parikh, Assistant Clinical Professor, Co-Assistant Director Interventional Cardiology Research, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 18-001544
Record Dates: First submitted 2022-05-09; First posted 2022-05-13 (Actual); Results first posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-02

CONDITIONS: Cardiac Allograft Vasculopathy
Keywords: Heart Transplantation; Endothelin-1; Cardiac Allograft Vasculopathy
MeSH Terms: interventions — macitentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Intervention Arm (Experimental): A consecutive subset of eligible patients based on inclusion/exclusion criteria will receive a 1-week course of Macitentan (10 mg po daily) prior to their routine 1-year coronary angiogram (7th and final dose of Macitentan will occur on the day of the angiogram).
  Interventions: Drug: Macitentan

INTERVENTIONS:
Drug: Macitentan — Macitentan is a nonselective endothelin-receptor antagonist (ERA) that is approved for use in pulmonary arterial hypertension (PAH); the use of Macitentan in post-heart transplant patients is considered investigational.
  Other Names: Opsumit

SUMMARY:
Many patients with end-stage heart failure, a condition in which the heart fails to pump enough blood to support the body's other organs, are fortunate enough to receive a heart transplant. However, despite taking medicines aimed at blunting the immune system's response to the donor heart, some of them will develop transplant-related disease in the coronary arteries supplying their hearts. Fifty years after the first human-to-human heart transplant, this disorder-cardiac allograft vasculopathy (CAV)-remains a leading cause of long-term death and has been coined the 'Achilles' Heel' of heart transplantation. Indeed, a better understanding of how CAV occurs and improved therapies to prevent and/or slow its development are desperately needed to meaningfully impact patient outcomes.

Endothelin-1 (ET-1) is a key molecular regulator of arterial health, and our prior data suggests that it is associated with accelerated CAV. In this particular study of recent heart transplant recipients, we are asking: Does ET-1 contribute to the coronary artery's capacity to dilate/constrict? To answer this question, during the cardiac catheterization at 1 year post-transplant (standard of care), we will measure blood levels of ET-1 and perform an invasive evaluation of coronary vasomotor function inn a consecutive subset of patients who will have received a 1-week course of the oral endothelin receptor antagonist (macitentan) prior this catheterization, which will allow us to test how much ET-1 contributes to coronary responsiveness.

The findings from this study may provide the necessary foundation to study whether endothelin receptor antagonists are able to effectively reduce the rate of accelerated CAV.

ELIGIBILITY:
Inclusion Criteria:

* 1) New heart transplant recipients already enrolled into a prospective cohort (parent) study
* 1a) Underwent baseline coronary angiography within the first 4 months of heart transplantation
* 1b) Have yet to complete 1-year coronary angiogram
* 2) ≥18 years old
* 3) Have a serum creatinine < 2.0 mg/dL (to minimize risk of contrast-induced nephropathy)
* 4) Able to provide informed written consent.

Exclusion Criteria:

* 1) Multi-organ transplant
* 2) Transplant-related complications and comorbidities that preclude the ability to safely perform an invasive coronary evaluation in the cardiac catheterization laboratory
* 3) Pregnant women due to possible fetal harm; all women of childbearing potential must have a negative pregnancy test within 1 week of starting Macitentan, and 30 days after completing the one-week course of Macitentan.
* 4) Patients who are taking potent CYP3A4 inhibitors (e.g. ketoconazole, ritonavir) as these drugs can expose one to higher levels of macitentan
* 5) Cirrhosis or baseline liver function tests (AST/ALT) > 3x the upper limit of normal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2022-05-19 (Actual); Primary Completion 2023-02-14 (Actual); Study Completion 2023-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rushi Parikh, MD, Principal Investigator — Assistant Clinical Professor; University of California, Los Angeles
Locations (1):
- Ronald Regan UCLA Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cooper DK. Christiaan Barnard and his contributions to heart transplantation. J Heart Lung Transplant. 2001 Jun;20(6):599-610. doi: 10.1016/s1053-2498(00)00245-x. PMID 11404164
- [Background] Lund LH, Edwards LB, Kucheryavaya AY, Benden C, Dipchand AI, Goldfarb S, Levvey BJ, Meiser B, Rossano JW, Yusen RD, Stehlik J. The Registry of the International Society for Heart and Lung Transplantation: Thirty-second Official Adult Heart Transplantation Report--2015; Focus Theme: Early Graft Failure. J Heart Lung Transplant. 2015 Oct;34(10):1244-54. doi: 10.1016/j.healun.2015.08.003. Epub 2015 Aug 28. No abstract available. PMID 26454738
- [Background] Chih S, Chong AY, Mielniczuk LM, Bhatt DL, Beanlands RS. Allograft Vasculopathy: The Achilles' Heel of Heart Transplantation. J Am Coll Cardiol. 2016 Jul 5;68(1):80-91. doi: 10.1016/j.jacc.2016.04.033. PMID 27364054
- [Background] Mitchell RN, Libby P. Vascular remodeling in transplant vasculopathy. Circ Res. 2007 Apr 13;100(7):967-78. doi: 10.1161/01.RES.0000261982.76892.09. PMID 17431198
- [Background] Kobashigawa JA, Tobis JM, Starling RC, Tuzcu EM, Smith AL, Valantine HA, Yeung AC, Mehra MR, Anzai H, Oeser BT, Abeywickrama KH, Murphy J, Cretin N. Multicenter intravascular ultrasound validation study among heart transplant recipients: outcomes after five years. J Am Coll Cardiol. 2005 May 3;45(9):1532-7. doi: 10.1016/j.jacc.2005.02.035. PMID 15862430
- [Background] Tuzcu EM, Kapadia SR, Sachar R, Ziada KM, Crowe TD, Feng J, Magyar WA, Hobbs RE, Starling RC, Young JB, McCarthy P, Nissen SE. Intravascular ultrasound evidence of angiographically silent progression in coronary atherosclerosis predicts long-term morbidity and mortality after cardiac transplantation. J Am Coll Cardiol. 2005 May 3;45(9):1538-42. doi: 10.1016/j.jacc.2004.12.076. PMID 15862431
- [Background] Bohm F, Pernow J. The importance of endothelin-1 for vascular dysfunction in cardiovascular disease. Cardiovasc Res. 2007 Oct 1;76(1):8-18. doi: 10.1016/j.cardiores.2007.06.004. Epub 2007 Jun 16. PMID 17617392
- [Background] Davenport AP, Hyndman KA, Dhaun N, Southan C, Kohan DE, Pollock JS, Pollock DM, Webb DJ, Maguire JJ. Endothelin. Pharmacol Rev. 2016 Apr;68(2):357-418. doi: 10.1124/pr.115.011833. PMID 26956245
- [Background] Sidharta PN, van Giersbergen PL, Dingemanse J. Safety, tolerability, pharmacokinetics, and pharmacodynamics of macitentan, an endothelin receptor antagonist, in an ascending multiple-dose study in healthy subjects. J Clin Pharmacol. 2013 Nov;53(11):1131-8. doi: 10.1002/jcph.152. Epub 2013 Sep 4. PMID 23900878
- [Background] Okada K, Nishida Y, Murakami H, Sugimoto I, Kosaka H, Morita H, Yamashita C, Okada M. Role of endogenous endothelin in the development of graft arteriosclerosis in rat cardiac allografts: antiproliferative effects of bosentan, a nonselective endothelin receptor antagonist. Circulation. 1998 Jun 16;97(23):2346-51. doi: 10.1161/01.cir.97.23.2346. PMID 9639379
- [Background] Simonson MS, Herman WH, Robinson A, Schulak J, Hricik DE. Inhibition of endothelin-converting enzyme attenuates transplant vasculopathy and rejection in rat cardiac allografts. Transplantation. 1999 Jun 27;67(12):1542-7. doi: 10.1097/00007890-199906270-00007. PMID 10401760
- [Background] Simonson MS, Robinson AV, Schulak JA, Hricik DE. Inhibition of endothelin-1 improves survival and vasculopathy in rat cardiac transplants treated with cyclosporine. Transplantation. 2002 Apr 15;73(7):1054-9. doi: 10.1097/00007890-200204150-00007. PMID 11965031
- [Background] Yamaguchi A, Miniati DN, Hirata Ki, Hoyt EG, Robbins RC. Ex vivo blockade of endothelin-1 inhibits graft coronary artery disease in a rodent cardiac allograft model. J Heart Lung Transplant. 2002 Apr;21(4):417-24. doi: 10.1016/s1053-2498(01)00397-7. PMID 11927217
- [Background] Ravalli S, Szabolcs M, Albala A, Michler RE, Cannon PJ. Increased immunoreactive endothelin-1 in human transplant coronary artery disease. Circulation. 1996 Nov 1;94(9):2096-102. doi: 10.1161/01.cir.94.9.2096. PMID 8901657
- [Background] Weis M, Wildhirt SM, Schulze C, Rieder G, Wilbert-Lampen U, Wolf WP, Arendt RM, Enders G, Meiser BM, von Scheidt W. Endothelin in coronary endothelial dysfunction early after human heart transplantation. J Heart Lung Transplant. 1999 Nov;18(11):1071-9. doi: 10.1016/s1053-2498(99)00081-9. PMID 10598730
- [Background] Ferri C, Properzi G, Tomassoni G, Santucci A, Desideri G, Giuliani AE, Starling RC, Ratliff NB, Cook DJ, McCarthy P, Young JB, Yamani MH. Patterns of myocardial endothelin-1 expression and outcome after cardiac transplantation. Circulation. 2002 Apr 16;105(15):1768-71. doi: 10.1161/01.cir.0000015606.69079.27. PMID 11956116
- [Background] Larose E, Behrendt D, Kinlay S, Selwyn AP, Ganz P, Fang JC. Endothelin-1 is a key mediator of coronary vasoconstriction in patients with transplant coronary arteriosclerosis. Circ Heart Fail. 2009 Sep;2(5):409-16. doi: 10.1161/CIRCHEARTFAILURE.108.836759. Epub 2009 Jun 15. PMID 19808370
- [Background] Starling RC, Stehlik J, Baran DA, Armstrong B, Stone JR, Ikle D, Morrison Y, Bridges ND, Putheti P, Strom TB, Bhasin M, Guleria I, Chandraker A, Sayegh M, Daly KP, Briscoe DM, Heeger PS; CTOT-05 consortium. Multicenter Analysis of Immune Biomarkers and Heart Transplant Outcomes: Results of the Clinical Trials in Organ Transplantation-05 Study. Am J Transplant. 2016 Jan;16(1):121-36. doi: 10.1111/ajt.13422. Epub 2015 Aug 10. PMID 26260101
- [Background] Pollack A, Nazif T, Mancini D, Weisz G. Detection and imaging of cardiac allograft vasculopathy. JACC Cardiovasc Imaging. 2013 May;6(5):613-23. doi: 10.1016/j.jcmg.2013.03.001. PMID 23680373
- [Background] Parikh RV, Khush K, Pargaonkar VS, Luikart H, Grimm D, Yu M, Okada K, Honda Y, Yeung AC, Valantine H, Fearon WF. Association of Endothelin-1 With Accelerated Cardiac Allograft Vasculopathy and Late Mortality Following Heart Transplantation. J Card Fail. 2019 Feb;25(2):97-104. doi: 10.1016/j.cardfail.2018.12.001. Epub 2018 Dec 10. PMID 30543947

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Arm
Started | 19
Completed | 17
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Intervention Arm
Number analyzed (Participants) | 19
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 54.2 [42.8 to 65.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 6
  Non-Hispanic White | 10
  Non-Hispanic Black | 1
  Non-Hispanic Asian | 1
  Other | 1
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Macitentan: Nitroglycerin (NTG) Luminal Dilation Ratio as Proportion of Vasomotor Tone Attributable to Endothelin-1 (ET-1)
Description: Macitentan: NTG luminal volume dilation ratio on Intravascular Ultrasound (IVUS). Vasodilation achieved by Macitentan was compared with that after intracoronary nitroglycerin, a maximal dilator of epicardial arteries, to determine the relative contribution of ET-1 to the overall resting vasomotor tone. The contribution of ET-1 to resting vasomotor tone is expressed as the ratio of dilation to Macitentan over the dilation to nitroglycerin.
Time Frame: End of study week 1 (time of 1 year post-transplant coronary angiogram)
Population: Sixteen patients had interpretable IVUS data.
Measure: Median (Inter-Quartile Range); unit: ratio
Groups:
- Participants With Progressive Cardiac Allograft Vasculopathy (CAV) at 1-year Post-transplant; Participants Without Progressive Cardiac Allograft Vasculopathy (CAV) at 1-year Post-transplant: A consecutive subset of eligible patients based on inclusion/exclusion criteria received a 1-week course of Macitentan (10 mg po daily) prior to their routine 1-year coronary angiogram (7th and final dose of Macitentan was on the day of the angiogram).
  Progressive CAV was defined as > 50th percentile of lumen volume loss measured by 3D IVUS
Arm/Group | Participants With Progressive Cardiac Allograft Vasculopathy (CAV) at 1-year Post-transplant | Participants Without Progressive Cardiac Allograft Vasculopathy (CAV) at 1-year Post-transplant
Number analyzed (Participants) | 8 | 8
ratio | 0.33 [0.31 to 0.37] | 0.30 [0.29 to 0.32]

ADVERSE EVENTS:
Time Frame: One week prior to one-year post-transplant angiogram (Day -7 to Study Day)
Arm/Group | Intervention Arm
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-28): https://cdn.clinicaltrials.gov/large-docs/08/NCT05373108/Prot_SAP_000.pdf